CLINICAL TRIAL: NCT03895242
Title: The Effect on Physiological Variables of Prone and Supine Positions Given to Preterm Infants Receiving Mechanical Ventilation
Brief Title: Prone and Supine Positions in Preterm Infants Receiving Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sultan Besiktas, Graduate Nurse, Akdeniz University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AkdenizU
Record Dates: First submitted 2019-03-24; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Preterm Infant; Ventilator Lung; Newborn; Preterm Birth
Keywords: Preterm infant; Mechanical ventilation; Position
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: The priority of the positions to be given to preterm infants was randomly determined.The positions of preterm infants was identified using the closed envelope method.The positions of infants were written in envelopes and closed.The clinical nurse, who was not in the research, pulled the envelope and identified the infant position.First group was first supine position,then prone position (n = 19), second group was first prone position, then supine position (n = 19).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:First supine position,then prone position (Experimental): First group was supine position then prone position.
  Interventions: Behavioral: Group 1:Supine-Prone
- Group 2:First prone position, then supine position (Experimental): Second group was first prone position, then supine position.
  Interventions: Behavioral: Group 2:Prone-Supine

INTERVENTIONS:
Behavioral: Group 1:Supine-Prone — After the infants were treated and fed, supine position was first given and waited for 60 minutes to stabilise (no data was collected during this time). After 61 minutes, it was allowed to stay in supine position for 2 hours. From the 61st minute, heart rate and oxygen saturation were evaluated in each infant in the supine positions at intervals of 15 min over a period of 120 min. At the end of two hours, the infant was given the prone position after the routine requirements such as diaper replacement were completed. Infants were waiting for 60 minutes to stabilize after the prone position (no data was collected during this time). From the 61st minute, heart rate and oxygen saturation were evaluated in each infant in the prone positions at intervals of 15 min over a period of 120 min.
  Arms: Group 1:First supine position,then prone position
Behavioral: Group 2:Prone-Supine — After the infants were treated and fed, prone position was first given and waited for 60 minutes to stabilise (no data was collected during this time). After 61 minutes, it was allowed to stay in prone position for 2 hours. From the 61st minute, heart rate and oxygen saturation were evaluated in each infant in the prone positions at intervals of 15 min over a period of 120 min. At the end of two hours, the infant was given the supine position after the routine requirements such as diaper replacement were completed. Infants were waiting for 60 minutes to stabilize after the supine position (no data was collected during this time). From the 61st minute, heart rate and oxygen saturation were evaluated in each infant in the prone positions at intervals of 15 min over a period of 120 min.
  Arms: Group 2:First prone position, then supine position

SUMMARY:
Positioning, which is one of the individualized developmental care methods, is known as the important care support process which is applied with the purpose of ensuring the least damage from the environmental. Positioning in preterm infants is the basis of neonatal nursing care. Positioning in preterm infants receiving mechanical ventilation support is important in terms of physiological and neurodevelopment. In infants undergoing respiratory support in NICU, it is important to determine the appropriate position, the frequency and duration of position change in order to reduce the oxygen need. In this respect, the aim of this study, designed as a randomized controlled trial, was to determine the effect of supine and prone positions on physiological variables (oxygen saturation and heart rate) of preterm infants receiving mechanical ventilation.

DETAILED DESCRIPTION:
In infants undergoing respiratory support in NICU, it is important to determine the appropriate position, the frequency and duration of position change in order to reduce the oxygen need. Therefore, the aim of this randomized controlled study, test the efficacy of two different positions (prone-supine) given to preterm newborns receiving mechanical ventilation.The study was conducted from February 2015 to June 2016.

Participants and setting:

We were interested in establishing the difference between the supine position and the prone position, with an error margin of 10%. According to the formula of the calculated sample size, for a crossover design with a = 0.05, the sample size required to achieve a 90% power is 36 infants. Thirty-eight infants who met the inclusion criteria of the study were selected and invited to participate. Of these, parents of 38 infants consented. A convenience sample of hospitalized preterm infants (less than 37 weeks gestational age) was selected from a tertiary neonatal intensive care unit of a teaching and research hospital in Turkey. Preterm infants were divided into two groups by randomization according to position priority (n = 38). First group was first supine position followed by prone position (n = 19), second group was first prone position, then supine position (n = 19). The priority of the positions to be given to preterm infants was randomly determined using the closed envelope method. The positions of infants were written in envelopes and closed. The clinical nurse, who was not in the research, pulled the envelope and identified position group of the infant . Thus, data were collected for both the prone and the supine position from a newborn.

Procedure and data collection:

The infants involved in the study were cared for in a incubator and wore diapers only. The temperature of the incubator was set to maintain a body temperature ranging from 36.5 to 37.2 °C. After necessary routine procedures such as diapering, body cleaning, weighing and suctioning were completed, each subject was randomly assigned to the supine-prone group or prone-supine group sequence. All of the positions of preterm infants were given carefully by the researcher.

Data Collection Tools:

Infant descriptive characteristics form: The form was developed in light of the relevant literature to collect data about gender, age, gestational age, body weight at study.

Infant's clinical variables form. The form was developed by the researchers according to the literature to collect data such as infant feeding method, caffeine and surfactant treatment.

Physiological variable monitoring form: The form was developed to record heart rate (HR) (min) and oxygen saturation (% SpO2) values in the literature.

Pulse Oximeter Device: A pulse oximetry was used to determine HR and SpO2. The physiological parameters were measured and recorded every 15 minute for a total of 120 minute. The normal vital sign ranges assumed for the study subjects were as follows; heart rate range of 121 to 179 beats per minute, oxygen saturation range ≥92%. The pulse oximetry was calibrated as recommended by the manufacturer prior to use at the beginning of each shift within the study period. The pulse oximetry probe was attached to the foot of the leg.All of the measurements were performed by researcher who carefully and prudently recorded the infants' response throughout the study process.

Positioning material:

Rolled sheets were used when infants were given positions.

Statistical analysis:

Data were analyzed using SPSS version 22.0 (SPSS Inc., Chicago, IL, USA) statistical program. Descriptive statistics were reported using frequencies, percentages, mean values, standard deviation, and range. The Kolmogorov-Smirnov test was conducted to assess the distribution of the variables in order to use a parametric or non-parametric test. All the variables were normally distributed. Therefore, parametric tests such as analysis of variance and t-test were used to determine the differences in variables between groups. Variance analysis was used for repeated measurements of heart rates and oxygen saturation measured by infants at 15 min intervals. A value of p <0.05 was considered statistically significant.

Ethical considerations:

İn the study, written consent was obtained from the ethics committee, institutions and families.

ELIGIBILITY:
Inclusion Criteria:

* Gestation week from 25 to 36 weeks
* Spontaneous breathing with mechanical ventilation (required ventilatory support and at least 12 hours in nasal continuous positive airway pressure therapy),
* Postnatal age ≤ 7 days,

Exclusion Criteria:

* Neuromuscular disease,
* Pulmonary arterial hypertension,
* Emphysema,
* Active bleeding,
* Respiratory problem due to heart disease,
* Obstacle to give birth position congenital disorder,
* Abdominal or thoracic surgery,
* Hypothermia and hyperthermia,
* Chest with tube,
* Continuous sedative treatment,
* Anticonvulsive therapy and cardiac drug therapy,
* Mechanical ventilator settings vary frequently,
* Preterm neonates with a frequency of more than three hours were not included in the study.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Heart Rate | An average of 2 year
  The number of heartbeats per minute was obtained using a pulse oximetry device. A separate pulse oximetry probe was inserted into each of the infants.
Oxygen Saturation | An average of 2 year
  Oxygen saturation (SpO2) was obtained using a pulse oximetry device. A separate pulse oximetry probe was inserted into each of the infants.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Study Director — Akdeniz University Children's Health and the Nursing Department; Sultan Beşiktaş, Principal Investigator — Antalya Health Sciences University Education and Research Hospital
Locations (1):
- Health Sciences University Education and Research Hospital, Neonatal Intensive Care Unit, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdeyazdan Z, Nematollahi M, Ghazavi Z, Mohhamadizadeh M. The effects of supine and prone positions on oxygenation in premature infants undergoing mechanical ventilation. Iran J Nurs Midwifery Res. 2010 Fall;15(4):229-33. PMID 22049286
- [Background] Chang YJ, Anderson GC, Dowling D, Lin CH. Decreased activity and oxygen desaturation in prone ventilated preterm infants during the first postnatal week. Heart Lung. 2002 Jan-Feb;31(1):34-42. doi: 10.1067/mhl.2002.120241. PMID 11805748